CLINICAL TRIAL: NCT05765188
Title: Impact of Age at Conization on Obstetrical Outcome: A Case-Control Study
Acronym: OBSTETRICON
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0049
Record Dates: First submitted 2018-09-17; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2018-09

CONDITIONS: Pregnancy Complications
Keywords: LEEP; preterm labor
MeSH Terms: conditions — Pregnancy Complications; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- < 25 years: 42 patients younger than 25 years at the time of loop electrosurgical excision procedure
  Interventions: Other: loop electrosurgical excision procedure
- > 25 years: 73 patients 25 years or older at the time of loop electrosurgical excision procedure
  Interventions: Other: loop electrosurgical excision procedure

INTERVENTIONS:
Other: loop electrosurgical excision procedure — A retrospective study of 115 women who underwent both loop electrosurgical excision procedure (LEEP) and subse- quent pregnancy follow-up in a referral center was conducted.

SUMMARY:
The maternity ward attached to the colposcopy clinic was also the obstetrical referral center for the region and carried out approximately 2500 deliveries per year. The aim of the study was to assess whether an age younger than 25 years at conization affected future pregnancy outcome as an independent factor. A retrospective study of 115 women who underwent both loop electrosurgical excision procedure (LEEP) and subsequent pregnancy follow-up in a referral center was conducted. Two groups were considered: patients younger than 25 years at the time of the loop electrosurgical excision procedure (n = 42) and 25 years or older (n = 73). Analyzed data were occurrence of preterm adverse obstetrical event and, specifically, preterm labor (PL) and preterm rupture of membranes; stratification based on term of occurrence was performed: less than 37 weeks of amenorrhea (WA), less than 34 WA, and less than 26 WA.

DETAILED DESCRIPTION:
The investigators conducted a retrospective observational study between January 2008 and December 2015 in a French colposcopic referral academic hospital. The maternity ward attached to the colposcopy clinic was also the obstetrical referral center for the region and carried out approximately 2500 deliveries per year. The aim of the study was to assess whether an age younger than 25 years at conization affected future pregnancy outcome as an independent factor. A retrospective study of 115 women who underwent both loop electrosurgical excision procedure (LEEP) and subsequent pregnancy follow-up in a referral center was conducted. Two groups were considered: patients younger than 25 years at the time of the loop electrosurgical excision procedure (n = 42) and 25 years or older (n = 73). Analyzed data were occurrence of preterm adverse obstetrical event and, specifically, preterm labor (PL) and preterm rupture of membranes; stratification based on term of occurrence was performed: less than 37 weeks of amenorrhea (WA), less than 34 WA, and less than 26 WA.

ELIGIBILITY:
Inclusion Criteria:

* female pregnant
* underwent loop electrosurgical excision procedure during the studied period
* delivered in their institution

Exclusion Criteria:

* patients having delivered elsewhere after loop electrosurgical excision procedure
* Early miscarriages (<14 weeks of amenorrhea )

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators recruited all patients who underwent loop electrosurgical excision procedure during the studied period and subsequently delivered in our institution. This only concerned the immediate after pregnancy: patients having delivered in our institution after having delivered elsewhere after loop electrosurgical excision procedure were excluded. Early miscarriages (<14 weeks of amenor- rhea [WA]) were also excluded. All patients were managed according to a multidisciplinary decision, based on French guidelines at the time of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
occurrence of preterm adverse obstetrical event in the group of women younger than < 25 years old | 18 weeks
  The objective of this study was to evaluate if an age younger than < 25 years old at the time of loop electrosurgical excision procedure affected future pregnancy and can have impact on th early preterm adverse obstetrical events.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Gondry, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No